CLINICAL TRIAL: NCT00543634
Title: Open-Label, Single-Dose, Partially Randomized, 6-Period, 6-Treatment, Crossover Bioavailability Study of 3 Pilot Formulations of Premarin®/Medroxyprogesterone Acetate (MPA) Compared With Reference Formulations of Premarin®/MPA (PREMPRO®) and MPA Suspension (Provera®) in Healthy Postmenopausal Women
Brief Title: Study Comparing Premarin®/MPA, PREMPRO® and Provera® in Healthy Postmenopausal Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Collaborators: MDS Pharma Services (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Wyeth
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 0713E1-1138
Record Dates: First submitted 2007-10-03; First posted 2007-10-15 (Estimated); Last update posted 2010-06-22 (Estimated); Status verified 2010-06

CONDITIONS: Postmenopause
MeSH Terms: interventions — Medroxyprogesterone Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: Premarin/MPA
- 2 (Active Comparator)
  Interventions: Drug: Provera 10 mg

INTERVENTIONS:
Drug: Premarin/MPA — 0.625 mg/2.5 mg X4
  Arms: 1
Drug: Premarin/MPA — 0.625 mg/5 mg X 2
  Arms: 1
Drug: Provera 10 mg — 2.5 mg of MPA, 4 tablets dissoved in water
  Arms: 2

SUMMARY:
The purpose of the study is to evaluate the safety and efficacy of new tablet formulations of Premarin®/medroxyprogesterone (MPA).

ELIGIBILITY:
* Healthy postmenopausal women aged 35 to 70 years with spontaneous or surgical amenorrhea
* BMI in the range of 18 to 35 kg/m2
* History or presence of hypertension (>139 mm Hg systolic or >89 mm Hg diastolic)
* History of drug allergy, particularly to conjugated estrogens (CE) or selective estrogen receptor modulators (SERMs)
* Use of any prescription or investigational drug within 30 days before test article administration

Ages: 35 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2007-10; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Plasma concentration data and pharmacokinetic (PK) parameters of MPA and Premarin® (estrone, equilin and MPA). | 4 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Omaha, Nebraska, United States